CLINICAL TRIAL: NCT02411422
Title: Comparison of Efficiency Between I-gel-Assisted Blind Intubation and I-gel-assisted Bronchoscopic Intubation During Cardiopulmonary Resuscitation: Randomized Simulation Study
Brief Title: Comparison of Efficiency Between I-gel Blind Intubation and I-gel Bronchoscopic Intubation During Resuscitation
Acronym: i-gel_br
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Choi Hyun Young, emergency medicine fellowship, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-02-30
Record Dates: First submitted 2015-03-18; First posted 2015-04-08 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Heart Arrest
Keywords: intubation; cardiopulmonary resuscitation; manikins
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intubation using laryngoscope (Experimental): Intubation using Macintosh laryngoscope. we will check procedure time according to kind of endotracheal tube, separately.
  Two kinds of endotracheal tube will be used
  * Conventional endotracheal tube
  * Reinforced endotracheal tube
  Interventions: Device: Conventional endotracheal tube; Device: Reinforced endotracheal tube
- i-gel blind intubation (Experimental): i-gel blind intubation means that blind endotracheal intubation will be performed after i-gel insertion.
  i-gel will be used as a conduit. we will check procedure time according to kind of endotracheal tube, separately.
  Two kinds of endotracheal tube will be used
  * Conventional endotracheal tube
  * Reinforced endotracheal tube
  Interventions: Device: Conventional endotracheal tube; Device: Reinforced endotracheal tube
- i-gel bronchoscopic intubation (Experimental): i-gel bronchoscopic intubation means that bronchoscopic endotracheal intubation will be performed after i-gel insertion.
  i-gel will be used as a conduit. we will check procedure time according to kind of endotracheal tube, separately.
  Two kinds of endotracheal tube will be used
  * Conventional endotracheal tube
  * Reinforced endotracheal tube
  Interventions: Device: Conventional endotracheal tube; Device: Reinforced endotracheal tube

INTERVENTIONS:
Device: Conventional endotracheal tube — Conventional endotracheal tube
Device: Reinforced endotracheal tube — Reinforced endotracheal tube

SUMMARY:
The investigators will compare conventional intubation using Macintosh laryngoscope, blind endotracheal intubation using i-gel for conduit and bronchoscopic intubation using Ambu-aScope and i-gel. All situation assumed as cardiac arrest. i.e, someone give chest compressions continuously without interruption.

Moreover the investigators will compare the type of endotracheal tube. Reinforced tube has more soft tube tip, so the investigators think it is more acceptable for intubation using i-gel as conduit.

ELIGIBILITY:
Inclusion Criteria:

* emergency physician
* work at emergency department more than 1 year.
* 50 or more experience of endotracheal intubation

Exclusion Criteria:

* having backache or wrist pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
intubation time | 1 Day
  1st intubation attempt, an expected average time is 1 min.

SECONDARY OUTCOMES:
success rate for intubation | 1 Day
  the rate for successful 1st intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sacred Heart Hospital, Seoul, Yeongdeungpo-gu, South Korea